CLINICAL TRIAL: NCT02987179
Title: Identification of Desaturation Episodes by Means of Continuous Measurement of Oxygen Saturation During Hemodialysis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Renal Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RRI-16-002
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: ESRD; Sleep Apnea; Oxygen Deficiency
MeSH Terms: conditions — Kidney Failure, Chronic; Sleep Apnea Syndromes; Hypoxia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ESRD Patients: The following inclusion criteria must be met for each subject.
  * Age ≥18 years and able to give written informed consent to the study
  * On chronic hemodialysis for ≥ 90 days at time of enrollment
  * Ability to read
  * Consent to have video recording taken during study visit
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Collect anthropomorphic, WatchPAT, Crit-line Monitor measurements as well as sleep questionnaires and video records

SUMMARY:
The clinical diagnosis of sleep apnea is difficult among ESRD patients since the characteristic clinical features of sleep apnea may be absent and since sleep-related symptoms, such as fatigue and sleepiness, may be attributed to kidney failure. However, the evaluation of patients with possible sleep apnea is the same among ESRD patients as in the general population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and able to give written informed consent to the study
* On chronic hemodialysis for ≥ 90 days at time of enrollment
* Ability to read
* Consent to have video recording taken during study visit

Exclusion Criteria:

* Subjects with cognitive impairment to consent
* Sickle cell anemia
* Prescription of nasal oxygen
* Simultaneous participation in another clinical trial that may affect breathing frequency/patterns, blood oxygenation, sleep/wake cycle or other parameters related to the outcomes of interest to this study
* Use of a breathing device, e.g. CPAP
* Central venous catheter used as vascular access for hemodialysis
* Artificial fingernails (may disturb the measurement of the WatchPAT)
* Use of one of the following medications: alpha blockers, short acting nitrates (less than 3 hours before the study).
* Permanent pacemaker
* Sustained non-sinus cardiac arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Identifying Intradialytis desaturation episodes | 1 week
  • To determine the sensitivity and specificity of the CLM for identifying intradialytic desaturation episodes, using the WatchPAT device as the reference method.

CONTACTS AND LOCATIONS:
Locations (1):
- Renal Research Institute, New York, New York, United States